CLINICAL TRIAL: NCT03084653
Title: Choosing the Technique for First Abdominal Entry in Laparoscopy: A Questionnaire-based Observational Study.
Brief Title: Choosing the Technique for First Abdominal Entry in Laparoscopy
Status: Completed | Type: Observational
Sponsor: Umraniye Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Fatih Basak, Medical Doctor, Umraniye Education and Research Hospital
Other Study IDs: Rationale-Trocar
Record Dates: First submitted 2017-03-09; First posted 2017-03-21 (Actual); Last update posted 2017-03-21 (Actual); Status verified 2017-03

CONDITIONS: Decision-Making
Keywords: Trocar entery; Surgery, Laparoscopic
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Survey: Close-ended survey questions were formed and will be sent to general surgeons by e-mail containing the web address of the survey.
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Close-ended survey will be performed to the participants. The survey consisted of 18 questions (Appendix). The first six questions (#1-6) were related with respondent's demographical and educational data and experiences of surgical and laparoscopic practices. There were five questions to determine preferred technique for first entry (#7-11), three questions for complications (#12-14), and remaining four questions for safety maneuvers (#15-18).

SUMMARY:
Several techniques for initial abdominal entry in laparoscopy have been introduced in literature. Various guidelines and recommendations are available on this subject, however, compliance to these are controversial. The purpose of this study is to evaluate the rationale and the process of decision making for first entry technique in laparoscopy.

DETAILED DESCRIPTION:
Several methods, i.e., the Veress needle, open approach using the Hasson trocar and direct trocar insertion without insufflation have been described for initial abdominal entry in laparoscopy. On the other hand, relatively new approaches, e.g., the optical or radially expanding trocars did not become common yet. Despite the advantages of laparoscopic surgery, serious complications can be encountered during the initial entry. Development of a complication, e.g., major vascular and intestinal injury, would affect the outcome of the operation and it may result in conversion to the open approach. Because of low incidence of these complications, it is impossible to show any superiority of one approach to another.

In this study, we aimed to analyze the rationale and the process of decision making of a surgeon about initial abdominal entry technique for laparoscopy.

ELIGIBILITY:
Inclusion Criteria:

* General Surgeons who approve to participate to the study will be included.

Exclusion Criteria:

* Surgical residents will be excluded from the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Close-ended survey questions were formed and sent to general surgeons by e-mail containing the web address of the survey.
Sampling Method: Non-Probability Sample
Enrollment: 263 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Rationale of choice in decision-making of first abdominal trocar entry method. | through study completion, an average of 1 year
  The survey will be performed to participant general surgeons to evaluate rationale of choice in decision-making of first abdominal trocar entry method.

CONTACTS AND LOCATIONS:
Overall Officials: Fatih Basak, Principal Investigator — Umraniye Education and Research Hospital
Locations (1):
- Umraniye Education and Research Hospital, Istanbul, Ümraniye, Turkey (Türkiye)